CLINICAL TRIAL: NCT00325130
Title: An Open-Label, Randomized, Multicenter Study of the Safety, Tolerability, and Immunogenicity of V501 Given Concomitantly With Menactra™ and ADACEL™ in Healthy Adolescents 11-17 Years of Age
Brief Title: Concomitant Use of Gardasil (V501) (Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine) With Combined Diphtheria, Tetanus, Pertussis Vaccine and Meningococcal Conjugate Vaccine in Adolescents (V501-025)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V501-025; 2005_092
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Results first posted 2009-07-13 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms, Glandular and Epithelial; Diphtheria; Tetanus; Whooping Cough; Meningitis
MeSH Terms: conditions — Neoplasms, Glandular and Epithelial; Diphtheria; Tetanus; Whooping Cough; Meningitis | interventions — Papillomavirus Vaccines; Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Concomitant Administration
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (HPV) vaccine; Biological: Comparator: Menactra™ (Concomitant); Biological: Comparator: Adacel™ (Concomitant)
- Group 2 (Experimental): Non-concomitant administration
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (HPV) vaccine; Biological: Comparator: Menactra™ (Non-concomitant); Biological: Comparator: Adacel™

INTERVENTIONS:
Biological: Comparator: Quadrivalent Human Papillomavirus (HPV) vaccine — Quadrivalent HPV vaccine was provided by the SPONSOR in single-dose vials containing a volume of 0.75 mL. The vaccine was administered as a
  0.5-mL intramuscular dose at Day 1, Month 2, and Month 6.
  Other Names: Gardasil
Biological: Comparator: Menactra™ (Concomitant) — A single administration of 0.5 mL intramuscular injection in a limb opposite that of quadrivalent HPV injection at Day 1
  Arms: Group 1
Biological: Comparator: Adacel™ (Concomitant) — a single administration of 0.5 mL intramuscular injection administered in a limb opposite that of quadrivalent HPV injection at Day 1
  Arms: Group 1
Biological: Comparator: Menactra™ (Non-concomitant) — A single administration of 0.5 mL intramuscular injection in a limb opposite that of quadrivalent HPV injection at Month 1
  Arms: Group 2
Biological: Comparator: Adacel™ — A single administration of 0.5 mL intramuscular injection in a limb opposite that of quadrivalent HPV injection at Month 1
  Arms: Group 2

SUMMARY:
Data from this study are expected to demonstrate that V501 (Human Papillomavirus (HPV) [Types 6, 11, 16, 18] Recombinant Vaccine) , when administered concomitantly with a combined diphtheria, tetanus, pertussis (Tdap) vaccine and a meningococcal conjugate vaccine in adolescents remains immunogenic and well-tolerated and it does not impair the immunogenicity of the concomitant vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy boys or girls, 11-17 years of age
* Must be a virgin with no intention of becoming sexually active during the study period
* Must have been properly vaccinated against diphtheria, tetanus and pertussis

Exclusion Criteria:

* Must not have received a vaccine against diphtheria, tetanus and pertussis in the past 5 years
* Must not have received any prior human papillomavirus (HPV) vaccine or meningococcal vaccine

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1042 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Reisinger KS, Block SL, Collins-Ogle M, Marchant C, Catlett M, Radley D, Sings HL, Haupt RM, Garner EI; Protocol 025 Investigators. Safety, tolerability, and immunogenicity of gardasil given concomitantly with Menactra and Adacel. Pediatrics. 2010 Jun;125(6):1142-51. doi: 10.1542/peds.2009-2336. Epub 2010 May 3. PMID 20439595

RESULTS

PARTICIPANT FLOW:
Groups:
- Concomitant Administration: Concomitant administration of quadrivalent HPV vaccine and Menactra™ and ADACEL™
- Non-concomitant Administration: Non-concomitant administration of quadrivalent HPV vaccine and Menactra™ and ADACEL™
Period: Overall Study
Arm/Group | Concomitant Administration | Non-concomitant Administration
Started | 518 | 524
Completed | 499 | 494
Not Completed | 19 | 30
Not completed — Lost to Follow-up | 6 | 14
Not completed — Withdrawal by Subject | 12 | 14
Not completed — Protocol Deviation | 0 | 1
Not completed — Moved | 0 | 1
Not completed — Patient Discontinued for Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Administration | Non-concomitant Administration | Total
Number analyzed (Participants) | 518 | 524 | 1042
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (1.84) | 12.7 (1.90) | 12.6 (1.88)
Age, Customized [Number; unit: participants]
  9 Years of Age and Under | 0 | 0 | 0
  10 to 17 Years of Age | 518 | 524 | 1042
  Over 17 Years of Age | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 340 | 648
  Male | 210 | 184 | 394
Race/Ethnicity [Number; unit: participants]
  Asian | 5 | 7 | 12
  Black | 54 | 74 | 128
  Hispanic American | 42 | 29 | 71
  Indian | 1 | 1 | 2
  Multi-Racial | 9 | 6 | 15
  Native American | 1 | 3 | 4
  White | 406 | 404 | 810

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Seroconverted for Human Papillomavirus (HPV) Type 6 (HPV 6 ≥ 20 mMU/mL) by Week 4 Postdose 3 (7 Months)
Time Frame: 7 Months
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 418 | 418
Participants | 416 | 417
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

2. Secondary Outcome: Acceptable Safety Profile
Time Frame: 15 days post injection
Reporting Status: Not Posted

3. Primary Outcome: Number of Subjects Who Seroconverted for HPV Type 11 (HPV 11 ≥ 16 mMU/mL) by Week 4 Postdose 3 (7 Months)
Time Frame: 7 Months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 418 | 418
Participants | 418 | 418
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

4. Primary Outcome: Number of Subjects Who Seroconverted for HPV Type 16 (HPV 16 ≥ 20 mMU/mL) by Week 4 Postdose 3 (7 Months)
Time Frame: 7 Months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 421 | 420
Participants | 421 | 420
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

5. Primary Outcome: Number of Subjects Who Seroconverted for HPV Type 18 (HPV 18≥ 24 mMU/mL) by Week 4 Postdose 3 (7 Months)
Time Frame: 7 Months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 423 | 421
Participants | 421 | 420
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -5%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

6. Primary Outcome: Number of Subjects Who Achieved a Four-fold Rise in Titers to Meningococcal Serogroup A One Month Postvaccination (Week 4 Postdose 1) With Menactra™
Time Frame: 7 Months
Population: Per-protocol population: subjects must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 424 | 412
Participants | 367 | 345
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

7. Primary Outcome: Number of Subjects Who Achieved a Four-fold Rise in Titers to Meningococcal Serogroup C One Month Postvaccination (Week 4 Postdose 1) With Menactra™
Time Frame: 7 Months
Population: Per-protocol population: subjects must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 451 | 422
Participants | 423 | 394
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

8. Primary Outcome: Number of Subjects Who Achieved a Four-fold Rise in Titers to Meningococcal Serogroup W-135 One Month Postvaccination (Week 4 Postdose 1) With Menactra™
Time Frame: 7 Months
Population: Per-protocol population: subjects must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 446 | 415
Participants | 429 | 394
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

9. Primary Outcome: Number of Subjects Who Achieved a Four-fold Rise in Titers to Meningococcal Serogroup Y One Month Postvaccination With Menactra™
Time Frame: 7 Months
Population: Per-protocol population: subjects must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 439 | 427
Participants | 414 | 404
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

10. Primary Outcome: Number of Subjects Who Achieved Acceptable Levels of Titers (Diphtheria ≥ 0.1 IU/mL) to Diphtheria One Month Postvaccination (Week 4 Postdose 1) With ADACEL™
Time Frame: 7 Months
Population: Per-protocol population: subjects must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 398 | 381
Participants | 397 | 381
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

11. Primary Outcome: Number of Subjects Who Achieved Acceptable Levels of Titers to Tetanus (Tetanus ≥ 0.1 IU/mL) One Month Postvaccination (Week 4 Postdose 1) With ADACEL™
Time Frame: 7 Months
Population: Per-protocol population: subjects must have no major protocol violations and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 398 | 384
Participants | 398 | 384
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The difference in seroconversion rates (concomitant group - nonconcomitant group) must be greater than -10%; p < 0.001, Miettinen & Nurminen — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; Miettinen & Nurminen method for difference in proportions, Stat Med 1985;4:213-26

12. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 6 at Week 4 Postdose 3 (7 Months) of GARDASIL™
Time Frame: 7 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 418 | 418
mMU/mL | 1349.3 [1189.7 to 1530.3] | 1340.8 [1181.6 to 1521.4]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

13. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 11 at Week 4 Postdose 3 (7 Months) of GARDASIL™
Time Frame: 7 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 418 | 418
mMU/mL | 1609.6 [1469.9 to 1762.6] | 1513.7 [1381.8 to 1658.1]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

14. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 16 at Week 4 Postdose 3 (7 Months) of GARDASIL™
Time Frame: 7 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 421 | 420
mMU/mL | 7203.0 [6448.0 to 8046.4] | 7370.0 [6593.6 to 8237.9]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

15. Primary Outcome: Geometric Mean Titers (GMTs) for Anti-HPV 18 at Week 4 Postdose 3 (7 Months) of GARDASIL™
Time Frame: 7 Months
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 423 | 421
mMU/mL | 1270.2 [1128.9 to 1429.1] | 1425.3 [1265.7 to 1605.1]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.5; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

16. Primary Outcome: Geometric Mean Titers (GMTs) for Pertussis Anti-Pertussis Toxin (Anti-PT) One Month Postvaccination (Week 4 Postdose 1) With ADACEL™
Time Frame: 7 Months
Population: Per-protocol population: subjects must
  have no major protocol violations and must have post-vaccination data.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 425 | 391
ELISA units/mL | 18.5 [16.9 to 20.2] | 19.3 [17.5 to 21.2]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

17. Primary Outcome: Geometric Mean Titers (GMTs) for Pertussis Anti-Filamentous Hemagglutinin) (Anti-FHA) One Month Postvaccination (Week 4 Postdose 1) With ADACEL™
Time Frame: 7 Months
Population: Per-protocol population: subjects must
  have no major protocol violations and must have post-vaccination data.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 430 | 402
ELISA units/mL | 132.5 [122.4 to 143.4] | 150.9 [138.9 to 164.0]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

18. Primary Outcome: Geometric Mean Titers (GMTs) for Pertussis Anti Pertactin (Anti-PRN) One Month Postvaccination (Week 4 Postdose 1) With ADACEL™
Time Frame: 7 Months
Population: Per-protocol population: subjects must
  have no major protocol violations and must have post-vaccination data.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 430 | 402
ELISA units/mL | 253.6 [229.8 to 279.9] | 274.2 [274.2 to 304.1]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

19. Primary Outcome: Geometric Mean Titers (GMTs) for Pertussis Anti-Fimbrial Agglutinogens 2/3 (Anti-FIM) One Month Postvaccination (Week 4 Postdose 1) With ADACEL™
Time Frame: 7 Months
Population: Per-protocol population: subjects must
  have no major protocol violations and must have post-vaccination data.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Concomitant Administration | Non-concomitant Administration
Number analyzed (Participants) | 430 | 402
ELISA units/mL | 703.0 [609.9 to 810.2] | 611.2 [526.4 to 709.6]
Statistical Analysis 1: Comparison: Concomitant Administration vs Non-concomitant Administration; Test type: Non-Inferiority or Equivalence — The ratio of GMTs (concomitant group / nonconcomitant group) must be greater than 0.67; p < 0.001, ANOVA — Since p<0.05, the hypothesis of noninferiority is accepted for this outcome; ANOVA on natural log titer with fixed effects for region, vaccination group and their interaction

ADVERSE EVENTS:
Arm/Group | Concomitant Administration | Non-concomitant Administration
Serious Adverse Events (participants affected / at risk) | 0 | 2
Other Adverse Events (participants affected / at risk) | 475 | 448
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Concomitant Administration | Non-concomitant Administration
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/522 | 1/498
Parotidectomy (General disorders) | 0/522 | 1/498
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Concomitant Administration | Non-concomitant Administration
Injection Site Pain quadrivalent HPV Vaccine postvaccination 1 (General disorders) | 315/514 | 228/406
Injection Site Swelling HPV Vaccine postvaccination 1 (General disorders) | 56/514 | 28/406
Injection Site Erythema qHPV Vaccine (postvaccination 2) (General disorders) | 53/506 | 61/492 — qHPV = quadrivalent HPV Vaccine
Injection Site Pain qHPV Vaccine (postvaccination 2) (General disorders) | 210/506 | 194/492
Injection Site Erythema qHPV Vaccine (postvaccination 3) (General disorders) | 68/503 | 60/485
Injection Site Pain qHPV Vaccine (postvaccination 3) (General disorders) | 253/503 | 234/485
Injection Site Swelling qHPV Vaccine (postvaccination 3) (General disorders) | 52/503 | 55/485
Injection Site Erythema ADACEL™ + Menactra™ (General disorders) | 121/514 | 107/401
Injection Site Pain ADACEL™ + Menactra™ (General disorders) | 421/514 | 303/401
Injection Site Swelling ADACEL™ + Menactra™ (General disorders) | 145/514 | 113/401
Headache Systemic Clinical (Nervous system disorders) | 113/520 | 114/498
Injection Site Erythema qHPV Vaccine (post-vaccination 1) (General disorders) | 37/514 | 26/406
Injection Site Swelling qHPV Vaccine (post-vaccination 2) (General disorders) | 42/506 | 48/492
Injection Site Bruising ADACEL™ + Menactra™ (General disorders) | 30/514 | 9/401
Abdominal Pain Upper (Gastrointestinal disorders) | 27/520 | 26/498
Pyrexia (General disorders) | 45/520 | 50/498
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 26/520 | 35/498

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.